CLINICAL TRIAL: NCT02807467
Title: Comparison of Propofol and Dexmedetomidine to Treat Hyperactive and Mixed ICU Delirium - the Basel ProDex Randomized Trial
Brief Title: Influence of Dexmedetomidine or Propofol on ICU Delirium
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: insufficient recruitment over a long period
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Basel ProDex Study
Record Dates: First submitted 2016-05-09; First posted 2016-06-21 (Estimated); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Delirium
Keywords: reduction; delirium; duration; severity
MeSH Terms: conditions — Delirium | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental): Dexmedetomidine is a potent selective α-2-adrenergic receptor agonist frequently used for sedation in the ICU, also among critically ill patients. It promotes sedation, anxiolysis, and moderate analgesia with minimal respiratory depression and has been shown to reduce severity and duration of ICU delirium.
  Interventions: Drug: Dexmedetomidine
- Propofol (Active Comparator): Standard therapy for ICU delirium.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — Continuous infusion of dexmedetomidine between 8pm and 6am after diagnosis of hyperactive or mixed delirium. The infusion might have to be repeated several times to achieve resolution of delirium.
  Other Names: Dexdor
  Arms: Dexmedetomidine
Drug: Propofol — Continuous infusion of propofol between 8pm and 6am after diagnosis of hyperactive or mixed delirium. The infusion might have to be repeated several times to achieve resolution of delirium.
  Other Names: Disoprivan
  Arms: Propofol

SUMMARY:
In this randomized study, the investigators aim to test the hypothesis that the reinstitution of a normal circadian rhythm by continuous infusions of dexmedetomidine compared to propofol between 8pm and 6am after diagnosis of hyperactive or mixed delirium, decreases the duration of delirium. The infusions might have to be repeated several times to achieve resolution of delirium.

DETAILED DESCRIPTION:
Dexmedetomidine is a potent selective α-2-adrenergic receptor agonist frequently used for sedation in the ICU, also among critically ill patients. It promotes sedation, anxiolysis, and moderate analgesia with minimal respiratory depression. Sedation of ICU patients remains challenging for doctors and nurses as there is evidence that the administration of sedatives in critically ill patients is potentially harmful mainly in relation to the delirium during critical care and the consecutive clinical outcome. However, in many cases, sedation is supportive for both patients and ICU personnel allowing controlled interactions with the patient through the established comfort and security, which upholds the patient's autonomy and herewith creates a less threatening environment. Delirium is frequent in acutely ill hospitalized patients, especially after cardiac or orthopaedic surgery, and in the ICU, and is associated with adverse outcome. It is a pathologic neurobehavioural syndrome caused by transient alteration of the normal neuronal network activity secondary to systemic disturbances. There is much effort to fight pain, agitation and delirium in the ICU where the majority of cases have to be dealt with. Many different sedatives are essential to calm the agitated or aggressive patients, despite the fact that sedatives bare the inherent risk of acute encephalopathy, especially in the post-sedation phase further aggravating the patient's status and thereby worsening outcome. However, the prognosis in patients with untreated ICU delirium is even worse.

In the surgical ICU of the University Hospital of Basel, standard therapy of delirium consists of the intravenous administration of haloperidol either parenteral or oral and oral quetiapine. At present, despite the recommendation against their use in the latest American guidelines for sedation, analgesia and delirium (Reference: College of Critical Care Medicine (CCM) Guidelines sedation, analgesia and delirium) and ongoing concern for its safety and efficacy, haloperidol is the first-line agent used worldwide for the treatment of delirium in general. However, there seems to be evidence for its potential to prevent delirium. Due to the disturbed circadian rhythm among delirious patients, exclusive sedation with haloperidol and quetiapine, especially at night, is insufficient frequently calling for additional sedative agents, such as propofol. There is evidence for beneficial effects on the circadian rhythm by dexmedetomidine which induces a unique sleep-like sedation state and in highly selected patients, dexmedetomidine infusions at night inducing light sedation could be shown to increase sleep efficiency and shift the 24h sleep pattern mainly to the night. The mechanism of action of dexmedetomidine is unique compared to traditionally administered sedative agents due to its lack of activity at the γ-aminobutyric acid receptor and missing anticholinergic activity. Mentioned side-effects of dexmedetomidine include bradycardia and hypotension with the need for vasoactive support in some cases.

The participants in this cohort will always have increased sympathetic tones, so hypotension and bradycardia are expected only in very few cases. Dexmedetomidine infusion is therefore not suggested for the treatment of acute agitation where bolus therapy is advised. There seems to be no negative effects on mortality but data suggest a highly significant reduction of incidence of delirium, agitation and confusion, lower treatment costs, reduction of ventilator days in less critically ill patients, and reduction of ICU and hospital stay when dexmedetomidine is used as a sedative agent. One study revealed that dexmedetomidine does not reduce the incidence but the duration of delirium; however, this study was restricted to postcardiotomy delirium. Another study measured a significant reduction of the incidence of postcardiotomy delirium, and one study in non-postcardiotomy patients also doubts the beneficial effect of dexmedetomidine in this context. These conflicting results call for further research in this field. Especially the role of dexmedetomidine in unique patient populations, such as neurosurgery, trauma and obstetrics still has to be evaluated but is not focused on in this investigation.

In this randomized study, the investigators aim to test the hypothesis that the reinstitution of a normal circadian rhythm by continuous infusions of dexmedetomidine compared to propofol between 8pm and 6am after diagnosis of hyperactive or mixed delirium, decreases the duration of delirium. The infusions might have to be repeated several times to achieve resolution of delirium.

For delirium assessment the investigators will follow the Intensive Care Delirium Screening Checklist (ICDSC) , for assessment of sedation level the investigators will comply with the Sedation Agitation Scale (SAS) and the Richmond Agitation Sedation Scale (RASS) , and for pain with the Critical care Pain Observational Tool (C-POT) and/or Visual Analogue Scale/Numeric Rating Scale (VAS/NRS) scales.

To evaluate potential side effects (see next section: study drugs) the investigators will record the following parameters:

* Fluid balance
* Blood count
* Creatinine
* Blood urea nitrogen
* Triglycerides Creatine kinase, myoglobin and lactate will be monitored to evaluate propofol related infusion Syndrome (PRIS), a threatening side effect of long-term propofol infusion. If the latter mentioned values are elevated the investigators would perform a muscle biopsy, for the syndrome leads to haemodynamic abnormalities, lactic acidosis and rhabdomyolysis.

The evaluation of the electroencephalogram (EEG) will enable the investigators to analyze different patterns of sleep architecture under the influence of dexmedetomidine and propofol. Interneuronal communication is based on electrical impulses and can be measured by EEG at any time, even during sleep.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 years or older) in a state of delirium (hyperactive ore mixed type) upon detection in the ICU (i.e., ICDSC >3).

Exclusion Criteria:

* Hypersensitivity to the active substance
* Advanced heart block (grade 2 or 3) unless implanted pacemaker
* Uncontrolled hypotension
* Severe cardiac dysfunction
* Bradycardia
* Egg allergy
* Soybean/soy allergy
* Age below 18 years
* Terminal state
* Pregnancy
* Active psychosis (of non organic origin = functional disturbances)
* Status epilepticus or postictal states following seizures on EEG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2023-02-11 (Actual)

PRIMARY OUTCOMES:
Reduction of ICU delirium duration assessed by ICDSC checklist | during stay at ICU, an average of 3 days; Delirium duration assessed every 8 hours starting with patient's ICU admission until delirium has subsided
  The onset of delirium will be defined as the start of the ﬁrst of a minimum of two subsequent shifts with an ICDSC ≥ 4 and an SAS ≥ 5. The end of the delirium will be defined as the end of the last shift with an ICDSC ≥ 4 that precedes a minimum of two subsequent shifts with an I CDSC < 4.

CONTACTS AND LOCATIONS:
Overall Officials: Alexa Hollinger, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Intensive Care Units, University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
anonymized data will be analyzed and published

REFERENCES:
- [Derived] Hollinger A, Ledergerber K, von Felten S, Sutter R, Ruegg S, Gantner L, Zimmermann S, Blum A, Steiner LA, Marsch S, Siegemund M. Comparison of propofol and dexmedetomidine infused overnight to treat hyperactive and mixed ICU delirium: a protocol for the Basel ProDex clinical trial. BMJ Open. 2017 Jul 13;7(7):e015783. doi: 10.1136/bmjopen-2016-015783. PMID 28710219